CLINICAL TRIAL: NCT03224624
Title: Self-management of Blood Pressure Medication for Hypertensive Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 15-369
Record Dates: First submitted 2017-07-11; First posted 2017-07-21 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either usual care or self-management of blood pressure using a stepped approach which participants can trigger using their home blood pressure measures.
Who Masked: Outcomes Assessor
Masking Description: The outcome (in clinic blood pressure) will be assessed without knowledge of which group participants were assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- self-management (Experimental): Participants will be taught to monitor blood pressure and make limited adjustments to their medications
  Interventions: Other: self-management protocol for hypertension care
- usual care (No Intervention): Participants will be enrolled in the study and undergo a baseline, 6 month, and 1 year visit but their hypertension care will be per usual care.

INTERVENTIONS:
Other: self-management protocol for hypertension care — participants in this arm will be taught to monitor and record their blood pressure. On a regular basis they will evaluate their blood pressure record and follow an algorithm to decide whether to adjust their medication.
  Arms: self-management

SUMMARY:
Hypertension is the most common medical problem among US Veterans. Treatment is available and effective, but control rates remain under 75%. While blood pressure control has traditionally been achieved through sequential visits and medication changes initiated by providers during office-based care, self-monitoring and self-management of blood pressure medication is an important strategy that would empower Veterans to achieve better control of blood pressure. The health impacts of better systems for treatment of hypertension are significant, including decreased rates of cardiovascular and kidney disease.

This two-site clinical trial will randomize 400 Veterans to either usual blood pressure care or a self-management strategy in which patient-driven self-management of blood pressure medications will be taught and used over the course of 1 year.

DETAILED DESCRIPTION:
Project background: Recent literature from the UK (TASMIN2 and TASMIN-SR trials) have suggested that patient-driven self-management of blood pressure medications can be effective in achieving hypertension control, but questions remain as to how to apply these findings to a US population. The VA Healthcare System is an ideal system in which to test and customize this strategy for blood pressure treatment.

Project question:

Is patient-initiated self-management of blood pressure medication using a pre-specified, generalizable dose escalation scheme clinically effective, safe, and acceptable to patients and clinicians, compared to usual care in controlling blood pressure in hypertensive Veterans? Project methods: The investigators propose a 12-month randomized, controlled, non-blinded, single-center study of patient-initiated self-management of blood pressure medication vs. usual care with planned post study cohort follow-up via medical records. Participants in the intervention arm will be provided with home blood pressure monitoring tools and a self-management algorithm for changing their blood pressure medications as needed. Participants in the usual care arm will receive home monitoring tools and typical hypertension care from the primary care provider. The primary blood pressure outcome measure for the study will be between-group change in in-clinic blood pressure. Acceptability, safety, patient-centered outcomes and adherence will be key secondary outcomes

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are those with who have a clinical diagnosis of hypertension
* Who are not currently at their in-clinic goal blood pressure (>130 or > 90 at minimum)
* Are able to provide independent informed consent and expected to be in the area for at least 12 months

Exclusion Criteria:

* Criteria for exclusion will include: active prescriptions for > 2 antihypertensive agents
* Known allergies to 2 or more antihypertensive agents
* Currently not primarily in charge of his/her own medication administration, e.g.:

  * those living in institutions or with dementia or other limitations making self medication care not possible
* Life expectancy of less than 12 months
* Blood pressure at screening visit > 180 mm Hg systolic or > 110 diastolic, or < 120 systolic
* Screening cognitive function (Montreal Assessment of Cognitive Function, MoCA) 48 score less than 25
* eGFR < 25 ml/min /1.73m2 or end-stage renal disease (ESRD)
* Inability to use a standard home blood pressure cuff
* Known secondary cause of hypertension that causes concern regarding safety of the protocol, in the opinion of the site investigator
* Cardiovascular event or hospitalization for unstable angina within last 3 months
* Symptomatic heart failure within the past 6 months or left ventricular ejection fraction < 35%
* Pregnancy or planned pregnancy, or of child-bearing age not using birth control
* Current participation in another clinical trial
* Or major factors judged to be likely to significantly limit comprehension of or adherence to interventions including:

  * dementia
  * psychiatric disease
  * substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dena Evette Rifkin, MD MS, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (2):
- United States (2):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
de-identified data may be shared at end of study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from opt-out letters, referrals, and advertisement. After consent, participants were assessed for eligibility by review of inclusion/exclusion criteria including BP at the screening visit as well as cognitive assessment.
Pre-assignment Details: Of 232 assessed, 111 did not randomize given inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | Self-management | Usual Care
Started | 60 | 61
Baseline Visit (Loss to in-person baseline visits due to COVID-19) | 59 | 60
6 Month Visit Completed (some 6 month visits modified to telephone or passive follow-up due to COVID-19) | 50 | 55
Completed (some 12 month visits completed as telephone or passive followup due to COVID-19) | 50 | 57
Not Completed | 10 | 4
Not completed — Lost to Follow-up | 9 | 4
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-management | Usual Care | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.5) | 63.3 (12.7) | 63.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 56 | 59 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 51 | 53 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 12 | 11 | 23
  White | 37 | 38 | 75
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59 | 60 | 119
Site [Count of Participants; unit: Participants]
  VA San Diego | 43 | 43 | 86
  VA San Francisco | 16 | 17 | 33
SBP at primary care visit [Mean (Standard Deviation); unit: mm Hg] | 147.0 (13.2) | 148.2 (11.5) | 147.59 (12.33)
DBP at primary care visit [Mean (Standard Deviation); unit: mm Hg] | 85.1 (8.4) | 82.7 (9.1) | 83.87 (8.81)
SBP at screening visit [Mean (Standard Deviation); unit: mm Hg] — Using standardized automated cuff and average of 2nd and 3rd reading.
  mm Hg | 141.9 (10.0) | 140.7 (8.9) | 141.29 (9.46)
DBP at screening visit [Mean (Standard Deviation); unit: mm Hg] | 83.7 (10.71) | 80.1 (12.9) | 81.89 (11.95)
alcohol use [Count of Participants; unit: Participants]
  current | 38 | 37 | 75
  former | 14 | 21 | 35
  never | 6 | 2 | 8
  unknown | 1 | 0 | 1
Smoking status [Count of Participants; unit: Participants]
  current | 6 | 3 | 9
  former | 24 | 28 | 52
  never | 29 | 29 | 58
Estimated GFR (creatinine-based) [Mean (Standard Deviation); unit: ml/min/1.73 M2 (CKD-EPI equation)] | 82.9 (19.0) | 78.5 (17.3) | 80.7 (18.2)
Duration of hypertension (years) [Mean (Standard Deviation); unit: years] | 13.2 (11.1) | 13.9 (11.6) | 13.5 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: In-clinic Blood Pressure Change
Description: Blood pressure as measured in clinic at start and end of study. **Due to COVID, a more limited number of participants were seen in person at end of study. Study protocol was modified to collect data by phone and via chart as well when in-person data collection was not feasible.
  Here, we report the strict definition and numbers seen in person as per the primary protocol.
Time Frame: baseline compared to 6 months (mid-study) and 1 year (end of intervention)
Population: Participants seen in person for blood pressure evaluation.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Self-management | Usual Care
Number analyzed (Participants) | 59 | 60
mm Hg
  mean SBP baseline | 136.0 (13.3) | 140.3 (12.4)
  mean SBP 12-month: number analyzed (Participants) | 37 | 42
  mean SBP 12-month | 126.9 (13.8) | 136.1 (12.2)
  difference in SBP baseline-12 month: number analyzed (Participants) | 37 | 42
  difference in SBP baseline-12 month | -6.95 (16.4) | -5.60 (17.6)
  mean DBP baseline | 80.5 (10.4) | 78.7 (13.1)
  mean DBP 12 month: number analyzed (Participants) | 37 | 42
  mean DBP 12 month | 73.4 (10.5) | 76.1 (13.1)
  DBP difference baseline-12 month: number analyzed (Participants) | 37 | 42
  DBP difference baseline-12 month | -5.51 (10.7) | -1.76 (12.0)
Statistical Analysis 1: Comparison: Self-management vs Usual Care; t- tests were done to compare group mean differences between self-management and usual care and within groups Mean differences were calculated by subtracting 12-month blood pressure from baseline blood pressure for each participant. t-tests were done to compare mean differences between the two groups; Test type: Equivalence — Comparing baseline->12month SBP change (mean difference) between the two groups; p = 0.72, t-test, 2 sided — p<0.05 considered significant; Mean Difference (Net) = -1.35, Standard Error of Mean 3.8 — direction of comparison: (self-management change over 12 months) - (usual care change over 12 months) in SBP
Statistical Analysis 2: Comparison: Self-management vs Usual Care; Mean differences were calculated by subtracting 12-month blood pressure from baseline blood pressure for each participant. t-tests were done to compare mean differences between the two groups; Test type: Equivalence — Comparing baseline->12month DBP change (mean difference) between the two groups; p = 0.15, t-test, 2 sided; Mean Difference (Net) = -3.75, Standard Error of Mean 2.55 — direction of comparison: (self-management change over 12 months) - (usual care change over 12 months) in DBP
Statistical Analysis 3: Comparison: Self-management; change in SBP from baseline to 12-months within self-management group; Test type: Equivalence — Comparing baseline->12month SBP change within self-management group (null hypothesis no change); p = 0.01, t-test, 2 sided; Mean Difference (Net) = -6.95 — (12-month SBP)-(baseline SBP) for self-management group (as given in table)
Statistical Analysis 4: Comparison: Usual Care; Comparing baseline->12month SBP change within usual care group; Test type: Equivalence — Comparing baseline->12month SBP change within usual care group (null hypothesis no change); p < 0.05, t-test, 2 sided; Mean Difference (Net) = -5.59 — (12-month SBP)-(baseline SBP) for usual care group (as given in table)
Statistical Analysis 5: Comparison: Self-management; change in DBP from baseline to 12-months within self-management group; Test type: Equivalence — Comparing baseline->12month DBP change within self-management group (null hypothesis no change); p < 0.01, t-test, 2 sided; Mean Difference (Net) = -5.51 — (12-month DBP)-(baseline DBP) for self-management group (as given in table)
Statistical Analysis 6: Comparison: Usual Care; Test type: Equivalence — change in DBP from baseline to 12-months within usual care group; p = 0.34, t-test, 2 sided; Mean Difference (Net) = -1.76 — (12-month DBP)-(baseline DBP) for usual care group (as given in table)

2. Other Pre Specified Outcome: Intervention Acceptability (Patient-reported)
Description: Acceptability of the intervention as measured by patient-reported scale of acceptability. On a scale from 1 to 10, how likely would you be to continue such a program? Please select a number. (0= very unlikely, 5 = average, 10 = likely)
Time Frame: 1 year
Population: Participants in the intervention arm who answered program evaluation question at end of study (not asked in control arm).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-management | Usual Care
Number analyzed (Participants) | 50 | 0
units on a scale | 7.74 (2.83) |

3. Other Pre Specified Outcome: Self-efficacy (Patient-reported)
Description: Patients will report their hypertension-specific self-efficacy on a scale that will be repeated at start and end of study. On a scale of 1-10 (very unconfident to very confident). "How confident are you that you can titrate or adjust your blood pressure?"
Time Frame: 1 year
Population: Everyone who completed 12 month questionnaire on self-efficacy in regard to blood pressure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-management | Usual Care
Number analyzed (Participants) | 47 | 54
score on a scale | 7.59 (2.74) | 5.04 (3.68)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of enrollment through the 12 month visit.
Description: Adverse event collection included adverse events of special interest, as reported below, regarding emergency department visits for problems potentially related to hypertension.
Arm/Group | Self-management | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/59 | 0/60
Serious Adverse Events (participants affected / at risk) | 14/59 | 12/60
Other Adverse Events (participants affected / at risk) | 3/59 | 5/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-management (N=59) | Usual Care (N=60)
Hospitalization (surgical, planned) (Surgical and medical procedures) | 2 (2) | 5 (5)
Infection requiring hospitalization (Infections and infestations) | 1 (1) | 3 (3) — 1 dental infection, 1 salmonella infection, 1 viral URI (usual care); 1 osteomyelitis (self-management)
Gastrointestinal disease requiring hospitalization (Gastrointestinal disorders) | 4 (4) | 1 (1) — 1 GI bleed (UC); 2 GI bleeds, 1 bowel obstruction, 1 Crohn's disease exacerbation (SM)
Diabetic ketoacidosis requiring hospitalization (Endocrine disorders) | 2 (2) | 0 (0)
pulmonary embolism requiring hospitalization (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
atrial fibrillation requiring hospitalization (Cardiac disorders) | 0 (0) | 1 (1)
Stroke requiring hospitalization (Cardiac disorders) | 1 (1) | 1 (1) — One stroke was fatal and is reported in all-cause mortality.
Psychiatric disease requiring hospitalization (Psychiatric disorders) | 1 (1) | 0 (0)
drug toxicity requiring hospitalization (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — carbamazepine toxicity
vertigo (BPPV) requiring hospitalization (Ear and labyrinth disorders) | 1 (1) | 0 (0)
injurious fall requiring hospitalization (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-management (N=59) | Usual Care (N=60)
Hypertension evaluted in emergency department (Cardiac disorders) | 1 (1) | 1 (1) — Adverse events of special interest for this study were emergency department visits related to blood pressure or cardiac symptoms.
Chest pain evaluated in emergency department (Cardiac disorders) | 2 (2) | 2 (2) — Includes chest pain deemed non-cardiac after evaluation
syncope evaluated in emergency department (Cardiac disorders) | 0 (0) | 1 (1)
Drug-associated angioedema, evaluated in emergency department (Immune system disorders) | 0 (0) | 1 (1) — related to lisinopril

LIMITATIONS AND CAVEATS:
Due to impact of COVID-19, recruitment was heavily impacted; repeated ambulatory blood pressure readings proved infeasible and that outcome is not available.

The investigators report here the strict per protocol analysis of in person blood pressures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT03224624/Prot_SAP_000.pdf